CLINICAL TRIAL: NCT01245959
Title: Prospective Randomized Trial Comparing Induction Chemotherapy Plus Concurrent Chemoradiotherapy With Concurrent Chemoradiotherapy in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Induction Chemotherapy in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fudan University (Other); West China Hospital (Other); Huazhong University of Science and Technology (Other); Peking University Cancer Hospital & Institute (Other); Zhejiang Cancer Hospital (Other); Central South University (Other); Jiangsu Cancer Institute & Hospital (Other); First People's Hospital of Foshan (Other); The Third Affiliated Hospital of Harbin Medical University (Other); Cancer Hospital of Guangxi Medical University (Other); Jiangxi Provincial Cancer Hospital (Other); Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jun Ma, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YP2010171
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; Concurrent chemoradiotherapy; Induction chemotherapy; Clinical trial
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Docetaxel; Cisplatin; Fluorouracil; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Induction chemotherapy and concurrent chemoradiotherapy (Experimental): Patients receive docetaxel (60mg/m2 on day 1), cisplatin (60mg/m2 on day 1) and fluorouracil (600mg/m2 on Days 1 to 5) every three weeks for three cycles before the radiotherapy, and then receive radical radiotherapy and cisplatin (100mg/m2) every three weeks for three cycles during radiotherapy.
  Interventions: Drug: Docetaxel, cisplatin and fluorouracil; Radiation: Concurrent chemoradiotherapy
- Concurrent chemoradiotherapy (Active Comparator): Patients receive radical radiotherapy and cisplatin (100mg/m2) every three weeks for three cycles during radiotherapy.
  Interventions: Radiation: Concurrent chemoradiotherapy

INTERVENTIONS:
Drug: Docetaxel, cisplatin and fluorouracil — Patients receive docetaxel (60mg/m2 on day 1), cisplatin (60mg/m2 on day 1) and fluorouracil (600mg/m2 on Days 1 to 5) every three weeks for three cycles before the radiotherapy.
  Other Names: TPF induction chemotherapy
  Arms: Induction chemotherapy and concurrent chemoradiotherapy
Radiation: Concurrent chemoradiotherapy — Patients receive radical radiotherapy and cisplatin (100mg/m2) every three weeks for three cycles during radiotherapy.
  Other Names: Radical radiotherapy and concurrent cisplatin

SUMMARY:
The purpose of this study is to compare induction chemotherapy (docetaxel+cisplatin+fluorouracil) plus concurrent chemoradiotherapy with concurrent chemoradiotherapy in patients with locoregionally advanced nasopharyngeal carcinoma (NPC), in order to confirm the value of induction chemotherapy in NPC patients.

DETAILED DESCRIPTION:
Patients presented with non-keratinizing NPC and stage T3-4N1M0/TxN2-3M0 are randomly assigned to receive induction chemotherapy (docetaxel+cisplatin+fluorouracil) plus concurrent chemoradiotherapy (investigational arm) or concurrent chemoradiotherapy (control arm). Patients in both arms receive radical radiotherapy, and cisplatin (100mg/m2) every three weeks for three cycles during radiotherapy. Patients in the investigational arm receive docetaxel(60mg/m2 on day 1), cisplatin (60mg/m2 on day 1) and fluorouracil (600mg/m2 on Days 1 to 5) every three weeks for three cycles before the radiotherapy. Patients are stratified according to the treatment centers and stage. The primary end point is failure-free survival (FFS). Secondary end points include overall survival (OS), distant failure-free survival (D-FFS), locoregional failure-free survival (LR-FFS), initial response rates after treatments and toxic effects. All efficacy analyses are conducted in the intention-to-treat population; the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing (according to World Health Organization (WHO) histologically type).
* Tumor staged as T3-4N1/N2-3 (according to the 7th American Joint Commission on Cancer edition).
* No evidence of distant metastasis (M0).
* Satisfactory performance status: Karnofsky scale (KPS) > 70.
* Adequate marrow: leucocyte count ≥4000/μL, hemoglobin ≥90g/L and platelet count ≥100000/μL.
* Normal liver function test: Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤2.5×ULN, and bilirubin ≤ULN.
* Adequate renal function: creatinine clearance ≥60 ml/min.
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
* Age ≥60 years or <18 years.
* Treatment with palliative intent.
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
* Pregnancy or lactation.
* History of previous radiotherapy (except for non-melanomatous skin cancers outside intended RT treatment volume).
* Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 476 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | 3-year
  Failure-free survival is calculated from the date of randomisation to the date of treatment failure or death from any cause, whichever is first.

SECONDARY OUTCOMES:
Overall survival | 3-year
  Overall survival is calculated from randomization to death from any cause.
Locoregional failure-free survival | 3-year
  The latency (ie, time from randomisation) to the first locoregional failure
Distant failure-free survival | 3-year
  The latency (ie, time from randomisation) to the first remote failure
The initial response rates after treatments | A week after completion of the last cycle of induction chemotherapy and 16 weeks after completion of radiotherapy
Toxic effects | During and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D., Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Cancer incidence in five continents. Volume VIII. IARC Sci Publ. 2002;(155):1-781. No abstract available. PMID 12812229
- [Background] Stephen B. Edge, David R. Byrd, Carolyn C. Compton, April G. Fritz, Frederick L. Greene, and Andy Trotti. AJCC Cancer Staging Manual. 7th ed. New York: Springer, 2009: 41-46.
- [Background] Lai SZ, Li WF, Chen L, Luo W, Chen YY, Liu LZ, Sun Y, Lin AH, Liu MZ, Ma J. How does intensity-modulated radiotherapy versus conventional two-dimensional radiotherapy influence the treatment results in nasopharyngeal carcinoma patients? Int J Radiat Oncol Biol Phys. 2011 Jul 1;80(3):661-8. doi: 10.1016/j.ijrobp.2010.03.024. Epub 2010 Jul 17. PMID 20643517
- [Background] Baujat B, Audry H, Bourhis J, Chan AT, Onat H, Chua DT, Kwong DL, Al-Sarraf M, Chi KH, Hareyama M, Leung SF, Thephamongkhol K, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy in locally advanced nasopharyngeal carcinoma: an individual patient data meta-analysis of eight randomized trials and 1753 patients. Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):47-56. doi: 10.1016/j.ijrobp.2005.06.037. PMID 16377415
- [Background] Vermorken JB, Remenar E, van Herpen C, Gorlia T, Mesia R, Degardin M, Stewart JS, Jelic S, Betka J, Preiss JH, van den Weyngaert D, Awada A, Cupissol D, Kienzer HR, Rey A, Desaunois I, Bernier J, Lefebvre JL; EORTC 24971/TAX 323 Study Group. Cisplatin, fluorouracil, and docetaxel in unresectable head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1695-704. doi: 10.1056/NEJMoa071028. PMID 17960012
- [Background] Posner MR, Hershock DM, Blajman CR, Mickiewicz E, Winquist E, Gorbounova V, Tjulandin S, Shin DM, Cullen K, Ervin TJ, Murphy BA, Raez LE, Cohen RB, Spaulding M, Tishler RB, Roth B, Viroglio Rdel C, Venkatesan V, Romanov I, Agarwala S, Harter KW, Dugan M, Cmelak A, Markoe AM, Read PW, Steinbrenner L, Colevas AD, Norris CM Jr, Haddad RI; TAX 324 Study Group. Cisplatin and fluorouracil alone or with docetaxel in head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1705-15. doi: 10.1056/NEJMoa070956. PMID 17960013
- [Background] Qin-Hua Zhang, Wei Luo, Qi-Chao Zhou, Zhan Yu, Jun Ma, Meng-Zhong Liu. TPF induction chemotherapy followed by intensity-modulated radiotherapy and concomitant chemotherapy for locoregionally advanced nasopharyngeal carcinoma. Chinese Journal of Cancer Prevention and Treatment 16(8): 625-628, 2009.
- [Background] Guo L, Lin HX, Xu M, Chen QY, Wang CT, Huang PY. Phase I study of TPF neoadjuvant chemotherapy followed by radical radiotherapy in advanced nasopharyngeal carcinoma. Chin J Cancer. 2010 Feb;29(2):136-9. doi: 10.5732/cjc.009.10367. PMID 20109339
- [Background] Friedman J, Furberg, C, DeMets D. Fundamentals of clinical trials. New York: Springer-Verlag; 1998.
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Cox JD, Stetz J, Pajak TF. Toxicity criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1341-6. doi: 10.1016/0360-3016(95)00060-C. No abstract available. PMID 7713792
- [Background] Chow, S.C., Shao, J., Wang, H. Sample Size Calculations in Clinical Research. New York: Marcel Dekker; 2003.
- [Derived] Dong D, Zhang F, Zhong LZ, Fang MJ, Huang CL, Yao JJ, Sun Y, Tian J, Ma J, Tang LL. Development and validation of a novel MR imaging predictor of response to induction chemotherapy in locoregionally advanced nasopharyngeal cancer: a randomized controlled trial substudy (NCT01245959). BMC Med. 2019 Oct 23;17(1):190. doi: 10.1186/s12916-019-1422-6. PMID 31640711
- [Derived] Zhang Y, Li WF, Liu X, Chen L, Sun R, Sun Y, Liu Q, Ma J. Nomogram to predict the benefit of additional induction chemotherapy to concurrent chemoradiotherapy in locoregionally advanced nasopharyngeal carcinoma: Analysis of a multicenter, phase III randomized trial. Radiother Oncol. 2018 Oct;129(1):18-22. doi: 10.1016/j.radonc.2017.12.002. Epub 2017 Dec 16. PMID 29258695
- [Derived] Li WF, Chen L, Sun Y, Ma J. Induction chemotherapy for locoregionally advanced nasopharyngeal carcinoma. Chin J Cancer. 2016 Nov 15;35(1):94. doi: 10.1186/s40880-016-0157-4. PMID 27846913
- [Derived] Sun Y, Li WF, Chen NY, Zhang N, Hu GQ, Xie FY, Sun Y, Chen XZ, Li JG, Zhu XD, Hu CS, Xu XY, Chen YY, Hu WH, Guo L, Mo HY, Chen L, Mao YP, Sun R, Ai P, Liang SB, Long GX, Zheng BM, Feng XL, Gong XC, Li L, Shen CY, Xu JY, Guo Y, Chen YM, Zhang F, Lin L, Tang LL, Liu MZ, Ma J. Induction chemotherapy plus concurrent chemoradiotherapy versus concurrent chemoradiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: a phase 3, multicentre, randomised controlled trial. Lancet Oncol. 2016 Nov;17(11):1509-1520. doi: 10.1016/S1470-2045(16)30410-7. Epub 2016 Sep 27. PMID 27686945